CLINICAL TRIAL: NCT02446249
Title: Open-Label, Dose-Escalation Study Evaluating the Safety of a Single Administration of an Adeno-Associated Virus Vector Encoding Human Aquaporin-1 to One Parotid Salivary Gland in Individuals With Irradiation-Induced Parotid Salivary Hypofunction
Brief Title: Safety of a Single Administration of AAV2hAQP1, an Adeno-Associated Viral Vector Encoding Human Aquaporin-1 to One Parotid Salivary Gland in People With Irradiation-Induced Parotid Salivary Hypofunction
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MeiraGTx, LLC (Industry)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150129; 15-D-0129 (Other: NIDCR)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Head and Neck Cancer; Radiation Induced Xerostomia; Salivary Hypofunction
Keywords: Gene Therapy; Xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm dose escalation (Experimental): single arm dose escalation
  Interventions: Biological: AAV2hAQP1

INTERVENTIONS:
Biological: AAV2hAQP1 — Infusion of gene therapy

SUMMARY:
Background:

- Radiation can cause the parotid salivary glands to make less saliva (dry mouth). This can cause problems like infections and tooth decay. Researchers hope a new drug can help people with dry mouth caused by radiation.

Objectives:

- To examine the safety of AAV2hAQP1 gene therapy. To see if the drug increases saliva in people whose parotid glands have had radiation.

Eligibility:

- People at least 18 years of age with a history of radiation therapy for head and neck cancer.

Design:

Participants will be screened in 2 visits with:

* medical history
* physical exam
* scans of the head, neck, and chest
* intravenous administration of glycopyrrolate to stop saliva
* saliva collections
* sialogram which is a procedure in which a substance is injected in the parotid gland and X-rays are taken.
* non-drug infusion
* a small piece of skin being taken

3-5-day hospital stay: Participants will receive the gene infusion. The AAV2hAQP1 will be in a solution in a syringe. It will be slowly pushed into the parotid gland through the parotid duct, an opening in the mouth near the second upper molar tooth.

10 outpatient visits over 3 years. These may include:

* repeats of selected screening tests, including saliva collection
* blood and urine tests
* oral and dental examinations
* head and neck exams, including the use of a thin scope to see the back of the throat
* questionnaires
* a small piece of parotid tissue being taken by either a small scope through the parotid duct or by a small needle guided by ultrasound
* scans of the head and neck. For some, contrast will be injected in a vein
* completion of a diary about how the participant feels between visits
* swabs of teeth and gums to assess the microbiome of the mouth

DETAILED DESCRIPTION:
The treatment of most head and neck cancer patients includes ionizing radiation (IR). Salivary glands in the IR field suffer irreversible damage. There is no conventional treatment available to correct this condition. Our research group has been developing an adeno-associated virus vector based on the hypothesis that this vector is capable of safely transferring the human aquaporin-1 (hAQP1) cDNA gene to parotid glands of adult patients with IR-induced salivary hypofunction, resulting in an elevated salivary output. Human AQP1 is a plasma membrane protein that facilitates water movement across lipid bilayers. Minipig studies have shown that the AAV2hAQP1 strategy for restoring salivary flow to IR-damaged salivary glands is effective without untoward effects after salivary gland delivery. As a proof of concept that AQP1 would restore saliva flow in a human population, we recently completed a phase 1 clinical trial (06-D-0206) using an Adenovirus-based vector encoding AQP1 to a single previously irradiated parotid gland in eleven patients using an open label, single dose, dose-escalation design. All patients tolerated vector delivery and study procedures well and positive objective and subjective responses were seen in five patients, all at doses <5.8 times10(9) vp/gland. At higher doses the patients possibly initiated an immune response to the vector and no improvement in gland function was observed. These findings have encouraged us to pursue studies with AAV2 based vectors, which have demonstrated lower immunogenicity and more stable expression compared with adenoviral vectors. The purpose of this clinical protocol is to test the safety of AAV2hAQP1, with some measures of efficacy, in adult patients with established IR-induced parotid gland hypofunction. The targeted tissue site for the AAV2hAQP1 vector in the proposed study is a single parotid gland. In this Phase 1 dose-escalation study, safety will be evaluated using conventional clinical and immunological parameters. The primary outcome measure for biological efficacy will be parotid gland salivary output.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age
  2. History of external beam radiation therapy for head and neck cancer, with a mean dose equal to or greater than 15 Gy to a parotid gland.
  3. Abnormal parotid gland function as judged by both absence of unstimulated parotid salivary flow and a stimulated parotid salivary flow in the targeted parotid gland >0 and <0.3 mL/min/gland after 2% citrate stimulation.
  4. No evidence of recurrence of primary malignancy by otolaryngology (ENT) assessment. Additionally, all patients must have been disease-free of head and neck cancer for at least 5 years, a status to be determined at pre-dose screening using negative clinical exams and PET and or CT imaging of the neck and chest. The anatomic subset of HPV positive oropharyngeal cancer may be enrolled after 2 years post completion of therapy.
  5. Willingness to practice the required birth control method ("barrier" contraception, condoms, diaphragm) until AAV2hAQP1 is no longer detectable in their serum or saliva.
  6. Women who cannot bear children (post-menopausal or due to a surgical intervention) also will be required to practice barrier birth control methods until AAV2hAQP1 is no longer detectable in their serum or saliva.
  7. Ability to stay at the NIH hospital for the period of time necessary to complete each on-site phase of the protocol (3-5 days).
  8. No history of allergies to any medications or agents to be used in this protocol.
  9. On stable medications (greater than or equal to 2 months) for any underlying medical conditions at time of vector administration.

EXCLUSION CRITERIA:

1. Pregnant or lactating women. Women of childbearing potential are required to have a negative serum pregnancy test at screening and a negative urine pregnancy test within 48 hours prior to gene infusion.
2. Any experimental therapy within 3 months.
3. Any active respiratory tract infection in the 3 weeks prior to day 1 of the protocol
4. Active infection that requires the use of intravenous antibiotics and does not resolve at least 1 week before Day 1.
5. Uncontrolled ischemic heart disease: unstable angina, evidence of active ischemic heart disease on ECG, congestive heart failure (left ventricular ejection fraction < 45% on MUGA or echo) or cardiomyopathy.
6. Asthma or chronic obstructive pulmonary disease requiring regular inhaled or systemic corticosteroids.
7. Individuals with a history of autoimmune diseases affecting salivary glands, including Sjogren's syndrome, lupus, scleroderma, type I diabetes, sarcoidosis, amyloidosis, and chronic graft versus host disease. Organ specific autoimmune conditions may be included if clinically stable.
8. Use of systemic immunosuppressive medications (,i.e., corticosteroids). Topical corticosteroids are allowed.
9. Malignancy, other than head and neck, within past 3 years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin or in situ cervical carcinoma.
10. Active infections including Epstein-Barr virus (EBV), cytomegalovirus (CMV), hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
11. WBC <3000/microL or ANC <1500/microL or Hgb <10.0 g/dL or platelets <100,000/microL or absolute lymphocyte count less than or equal to 500/microL.
12. ALT and/or AST > 1.5 times upper limit of normal (ULN) or alkaline phosphatase >1.5 times ULN
13. Serum creatinine > 2 mg/dL.
14. Serum bilirubin measurements (total, direct, indirect) that are outside of the normal range.
15. Individuals who are active cigarette smokers as determined by self-reporting.
16. Individuals who have an allergy to iodine or shellfish and thus are unable to have sialographic evaluations.
17. Individuals who have an allergy or hypersensitivity to glycopyrrolate
18. Individuals whose parotid duct(s) are not clinically accessible on screening sialography.
19. Individuals, who on sialography, have a distal stenosis that would impede vector delivery and, for the expansion cohort, those who have a parotid volume >2.5 mL.
20. Significant concurrent or recently diagnosed (<2 months) medical condition that, in the opinion of the Medically Responsible Investigator, could affect the patient's ability to tolerate or complete the study.
21. Live vaccines within 4 weeks of first infusion.
22. Individuals who have had an adverse response to prednisone (i.e. hallucinations).
23. Individuals with uncontrolled diabetes (HbA1c greater than 10%).
24. Individuals with untreated severe dental caries, pyorrhea, gingivitis, chronic radiation mucositis or ulceration, erythroplasia, leukoplakia or other pre-malignant conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05-04; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety of vector | 36 months

SECONDARY OUTCOMES:
Efficacy of treatment | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: John A Chiorini, Ph.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gao R, Yan X, Zheng C, Goldsmith CM, Afione S, Hai B, Xu J, Zhou J, Zhang C, Chiorini JA, Baum BJ, Wang S. AAV2-mediated transfer of the human aquaporin-1 cDNA restores fluid secretion from irradiated miniature pig parotid glands. Gene Ther. 2011 Jan;18(1):38-42. doi: 10.1038/gt.2010.128. Epub 2010 Sep 30. PMID 20882054
- [Background] Baum BJ, Alevizos I, Zheng C, Cotrim AP, Liu S, McCullagh L, Goldsmith CM, Burbelo PD, Citrin DE, Mitchell JB, Nottingham LK, Rudy SF, Van Waes C, Whatley MA, Brahim JS, Chiorini JA, Danielides S, Turner RJ, Patronas NJ, Chen CC, Nikolov NP, Illei GG. Early responses to adenoviral-mediated transfer of the aquaporin-1 cDNA for radiation-induced salivary hypofunction. Proc Natl Acad Sci U S A. 2012 Nov 20;109(47):19403-7. doi: 10.1073/pnas.1210662109. Epub 2012 Nov 5. PMID 23129637
- [Background] Delporte C, O'Connell BC, He X, Lancaster HE, O'Connell AC, Agre P, Baum BJ. Increased fluid secretion after adenoviral-mediated transfer of the aquaporin-1 cDNA to irradiated rat salivary glands. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):3268-73. doi: 10.1073/pnas.94.7.3268. PMID 9096382
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-D-0129.html